CLINICAL TRIAL: NCT02136524
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE, RANDOMIZED, 2-PERIOD, 2-TREATMENT SEQUENCE CROSS-OVER STUDY TO ASSESS THE RELATIVE BIOAVAILABILITY OF COBIMETINIB ADMINISTERED AS A TABLET FORMULATION COMPARED TO A CAPSULE FORMULATION IN HEALTHY SUBJECTS
Brief Title: A Randomized, Phase I, Cross-Over Study to Assess the Relative Bioavailability of Single-Dose Cobimetinib (GDC-0973) in Tablet vs. Capsule Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: GP28370
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — cobimetinib

ARMS (2):
- Capsule formulation (Experimental)
  Interventions: Drug: cobimetinib
- Tablet formulation (Experimental)
  Interventions: Drug: cobimetinib

INTERVENTIONS:
Drug: cobimetinib — Single, oral dose given as a tablet on Day 1 after a minimum 8 h fast
  Other Names: GDC-0973, XL-518
  Arms: Tablet formulation
Drug: cobimetinib — Single, oral dose given as 4 capsules on Day 1 after a minimum 8 h fast
  Other Names: GDC-0973, XL-518
  Arms: Capsule formulation

SUMMARY:
This study will be a Phase 1, open-label, randomized, 2-period, 2-treatment sequence crossover study to determine the relative bioavailability of cobimetinib administered as a single dose of the tablet formulation relative to a single dose of the capsule formulation to healthy male and female participants. A minimum of 24 participants (12 participants per sequence) will complete the study. Participants will be randomly assigned to 2 possible sequences (i.e., I: A/B, II: B/A) where the treatments are as follows: Treatment A: One cobimetinib tablet administered as a single oral dose after at least an 8-hour fast; Treatment B: Four cobimetinib capsules administered as a single oral dose after at least an 8-hour fast. The study is expected to last approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers between 18 and 55 years of age, inclusive
* Body mass index between 18.5 to 32.0 kg/m2, inclusive;
* Adequate renal, liver, and hematologic function
* Participants who are in good health as determined by no clinically significant findings from medical history, 12-lead ECG, vital signs, and clinical laboratory evaluations

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Days 1 to 10 and 15 to 25 (1 to 10 of the second crossover sequence)
Time to maximum concentration (tmax) | Days 1 to 10 and 15 to 25 (1 to 10 of the second crossover sequence)
Area under the concentration-time curve (AUC) | Days 1 to 10 and 15 to 25 (1 to 10 of the second crossover sequence)
Apparent terminal elimination rate constant | Days 1 to 10 and 15 to 25 (1 to 10 of the second crossover sequence)
Half-life (t1/2) | Days 1 to 10 and 15 to 25 (1 to 10 of the second crossover sequence)
Apparent clearance (CL/F) | Days 1 to 10 and 15 to 25 (1 to 10 of the second crossover sequence)
Apparent volume of distribution (Vz/F) | Days 1 to 10 and 15 to 25 (1 to 10 of the second crossover sequence)
Relative bioavailability (Frel) | Days 1 to 10 and 15 to 25 (1 to 10 of the second crossover sequence)

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Dallas, Texas, United States